CLINICAL TRIAL: NCT02778100
Title: A Phase 1 Study to Evaluate the Effects of Common Cold and of Concomitant Administration of Nasal Decongestant on the Pharmacokinetics and Pharmacodynamics of a Novel Glucagon Formulation in Otherwise Healthy Subjects
Brief Title: A Study of Nasal Glucagon in Participants With a Common Cold
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Locemia Solutions ULC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16425; GUO-P2-628 (Other: AMG Medical Inc.); AMG 104 (Other: AMG Medical Inc.); I8R-MC-IGBE (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-05-18; First posted 2016-05-19 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2016-05

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold | interventions — Oxymetazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nasal Glucagon (NG) - Common Cold (Experimental): Cohort 1 - Nasal Glucagon (NG) administered once in participants with a common cold.
  Interventions: Drug: Nasal Glucagon
- Nasal Glucagon (NG) - Symptom-Free (Experimental): Cohort 1 - NG administered once in participants who have recovered from a common cold.
  Interventions: Drug: Nasal Glucagon
- NG - Common Cold+Oxymetazoline (Experimental): Cohort 2 - NG administered once in participants with a common cold who are taking oxymetazoline.
  Interventions: Drug: Nasal Glucagon; Drug: Oxymetazoline

INTERVENTIONS:
Drug: Nasal Glucagon — Administered intranasally.
  Other Names: LY900018; AMG 504-1
Drug: Oxymetazoline — Administered intranasally.
  Arms: NG - Common Cold+Oxymetazoline

SUMMARY:
The main purpose of this study is to evaluate the safety of nasal glucagon (NG) in participants with a common cold, some of whom will also take a nasal decongestant. The study will investigate how the body processes NG and the effect of NG on the body. The study will last up to 30 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant presenting a score of 2 or 3 on nasal congestion and/or nasal discharge associated with at least one other symptom of common cold, as determined by the 8-item Jackson cold scale at screening and prior to dosing of period 1.
* Participant with a body mass index (BMI) greater than or equal to 18.50 and below 30.00 kilogram per square meter (kg/m²).
* Light-, non- or ex-smokers.
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, biochemistry, electrocardiogram [ECG] and urinalysis).

Exclusion Criteria:

* Presence of any nose piercings.
* History of significant hypersensitivity to glucagon, oxymetazoline or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
* Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease.
* Presence of severe fever (more than 39.5 degrees Celsius) at screening or prior to dosing of period 1.
* Presence of clinically significant findings on nasal examination or bilateral anterior rhinoscopy, such as structural abnormalities, nasal polyps, marked septal deviation, nasal tumors.
* Presence or history of Type 1 or Type 2 diabetes.
* Presence or history of significant hypoglycemia or hyperglycemia.
* Use of beta-blockers, indomethacin, warfarin or anticholinergic drugs in the previous 28 days before day 1 of the study.
* Fasting blood glucose above 6.1 mmol/L at screening, following a 12-hour fasting period.
* Fasting blood glucose assessed with a glucose meter above 6.1 mmol/L approximately 0.5 hour before each dosing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Royal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Nasal Glucagon (NG) 3 mg (Milligram): Period 1:
  NG administered once in participants with a common cold.
  Period 2: NG administered once in participants who have recovered from a common cold.
- NG 3 mg Plus Oxymetazoline: Period 1 only: NG administered once to participants with a common cold, who are taking oxymetazoline.
Period: Period 1 (Common Cold)
Arm/Group | Nasal Glucagon (NG) 3 mg (Milligram) | NG 3 mg Plus Oxymetazoline
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2 (No Cold Symptoms)
Arm/Group | Nasal Glucagon (NG) 3 mg (Milligram) | NG 3 mg Plus Oxymetazoline
Started | 17 | 0 (Cohort 2 only administered NG to participants with a common cold who are taking oxymetazoline.)
Completed | 17 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled in Period 1.
Groups:
- Nasal Glucagon (NG): Dose of 3 mg NG administered once to participants with a common cold.
- NG Plus Oxymetazoline: Dose of 3 mg NG administered once to participants with a common cold, who are taking oxymetazoline.
- Total: Total of all reporting groups
Arm/Group | Nasal Glucagon (NG) | NG Plus Oxymetazoline | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 32 [20 to 50] | 29 [20 to 46] | 30.5 [20 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 2 | 3 | 5
  White | 16 | 14 | 30
  Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs)
Description: Safety and tolerability evaluated through the assessment of adverse events.
  A SAE (serious adverse event) was defined as any untoward medical occurrence in a clinical investigation participant administered the investigational product and which did not necessarily have a causal relationship with this treatment.
  A summary of other non-serious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline up to Study Completion (Day 30)
Population: All enrolled participants.
Measure: Count of Participants; unit: Participants
Groups:
- NG - Common Cold: Dose of 3 mg NG administered once in participants with a common cold.
- NG - Symptom-Free: Dose of 3 mg NG administered once in participants who have recovered from a common cold.
- NG - Common Cold+Oxymetazoline: Dose of 3 mg NG administered once in participants with a common cold who are taking oxymetazoline.
Arm/Group | NG - Common Cold | NG - Symptom-Free | NG - Common Cold+Oxymetazoline
Number analyzed (Participants) | 18 | 17 | 18
Participants | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to T (AUC[0-tlast]) of Baseline Adjusted Glucagon
Time Frame: Pre-dose; 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2.0, 2.5 and 3.0 hours after glucagon administration
Population: All enrolled participants with evaluable PK data.
Measure: Mean (Standard Deviation); unit: picogram*hour per millilitre (pg*hr/mL)
Arm/Group | NG - Common Cold | NG - Symptom-Free | NG - Common Cold+Oxymetazoline
Number analyzed (Participants) | 18 | 17 | 18
picogram*hour per millilitre (pg*hr/mL) | 1039.7 (1020.81) | 631.8 (399.66) | 868.4 (622.39)

3. Secondary Outcome: PK: Area Under the Curve Extrapolated to Infinity (AUC[0-inf]) of Baseline Adjusted Glucagon
Time Frame: Pre-dose; 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2.0, 2.5 and 3.0 hours after glucagon administration
Population: All enrolled participants with evaluable PK data.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | NG - Common Cold | NG - Symptom-Free | NG - Common Cold+Oxymetazoline
Number analyzed (Participants) | 18 | 17 | 18
pg*hr/mL | 1108.9 (1055) | 669.3 (431.7) | 1064.3 (838.4)

4. Secondary Outcome: PK: Time to Maximum Concentration (Tmax) of Baseline Adjusted Glucagon
Time Frame: Pre-dose; 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2.0, 2.5 and 3.0 hours after glucagon administration
Population: All enrolled participants with evaluable PK data.
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | NG - Common Cold | NG - Symptom-Free | NG - Common Cold+Oxymetazoline
Number analyzed (Participants) | 18 | 17 | 18
Hour (hr) | 0.3 [0.08 to 1.5] | 0.3 [0.25 to 0.67] | 0.3 [0.17 to 1.00]

5. Secondary Outcome: PK: Maximum Change From Baseline Concentration (Cmax) of Glucagon
Time Frame: Pre-dose; 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2.0, 2.5 and 3.0 hours after glucagon administration
Population: All enrolled participants with evaluable PK data.
Measure: Mean (Standard Deviation); unit: picograms per millilitre (pg/mL)
Arm/Group | NG - Common Cold | NG - Symptom-Free | NG - Common Cold+Oxymetazoline
Number analyzed (Participants) | 18 | 17 | 18
picograms per millilitre (pg/mL) | 1145.4 (994.43) | 745.6 (548.42) | 811.5 (597.51)

6. Secondary Outcome: Pharmacodynamics (PD): Area Under the Effect Concentration Time Curve (AUEC0-3) of Baseline-Adjusted Glucose From Time Zero up to 3 Hours
Time Frame: Pre-dose; 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2.0, 2.5 and 3.0 hours after glucagon administration
Population: All enrolled participants with evaluable PD data.
Measure: Mean (Standard Deviation); unit: Hour*millimoles per liter(hr*mmol/L)
Arm/Group | NG - Common Cold | NG - Symptom-Free | NG - Common Cold+Oxymetazoline
Number analyzed (Participants) | 18 | 17 | 18
Hour*millimoles per liter(hr*mmol/L) | 4.3 (2.11) | 3.8 (1.92) | 4.2 (2.06)

7. Secondary Outcome: PD: Time to Maximum Concentration (Tmax) of Baseline-Adjusted Glucose
Time Frame: Pre-dose; 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2.0, 2.5 and 3.0 hours after glucagon administration
Population: All enrolled participants with evaluable PD data.
Measure: Median (Full Range); unit: Millimoles per liter (mmol/L)
Arm/Group | NG - Common Cold | NG - Symptom-Free | NG - Common Cold+Oxymetazoline
Number analyzed (Participants) | 18 | 17 | 18
Millimoles per liter (mmol/L) | 0.5 [0.25 to 1.0] | 0.6 [0.33 to 1.00] | 0.7 [0.33 to 1.00]

8. Secondary Outcome: PD: Baseline-Adjusted Glucose Maximum Concentration (BGmax) of Baseline-Adjusted Glucose
Time Frame: Pre-dose; 0.08, 0.17, 0.25, 0.33, 0.5, 0.67, 1.0, 1.5, 2.0, 2.5 and 3.0 hours after glucagon administration
Population: All enrolled participants with evaluable PD data.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | NG - Common Cold | NG - Symptom-Free | NG - Common Cold+Oxymetazoline
Number analyzed (Participants) | 18 | 17 | 18
Millimoles per liter (mmol/L) | 2.9 (1.57) | 2.7 (1.38) | 3.4 (1.42)

ADVERSE EVENTS:
Time Frame: First dose of study drug (Day 1) until post-study completion (Day 30).
Groups:
- NG- Common Cold: Dose of 3 mg nasal glucagon (NG) administered once in participants with a common cold.
- NG - Symptom-Free: Dose of 3 mg nasal glucagon (NG) administered once in participants who have recovered from a common cold.
- NG - Common Cold+Oxymetazoline: Dose of 3 mg nasal glucagon (NG) administered once in participants with a common cold who are taking oxymetazoline.
Arm/Group | NG- Common Cold | NG - Symptom-Free | NG - Common Cold+Oxymetazoline
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 18/18 | 17/17 | 18/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NG- Common Cold (N=18) | NG - Symptom-Free (N=17) | NG - Common Cold+Oxymetazoline (N=18)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Eye pruritus (Eye disorders) | 5 (5) | 0 (0) | 5 (5)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 13 (17) | 12 (13) | 12 (16)
Ocular hyperaemia (Eye disorders) | 7 (7) | 7 (7) | 8 (12)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (10) | 2 (2) | 7 (7)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 5 (7)
Administration site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 2 (2) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sensation of pressure (General disorders) | 0 (0) | 0 (0) | 2 (2)
Administration related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 5 (6) | 5 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 5 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 6 (6) | 3 (3) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Self-induced vomiting (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 4 (4)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 7 (7) | 15 (15)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 5 (6) | 14 (15)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days